CLINICAL TRIAL: NCT06419179
Title: A Multicenter Phase II Trial of Maintenance Durvalumab (MEDI4736) and Olaparib (AZD2281) After Standard 1st Line Treatment (Carboplatin/Cisplatin, Etoposide, Durvalumab) in Homologous Recombination Deficiency (HRD) Positive Extensive Disease (ED) Small-cell Lung Cancer (SCLC)
Brief Title: Maintenance Durvalumab (MEDI4736) and Olaparib (AZD2281) After Standard 1st Line Treatment (Carboplatin/Cisplatin, Etoposide, Durvalumab) in HRD Positive Extensive Disease (ED) Small-cell Lung Cancer (SCLC)
Acronym: GUIDANCE
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Juergen Wolf, Clinical Prof. Dr. Jürgen Wolf, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-5159; 2024-512373-27-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-03; First posted 2024-05-17 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination of olaparib and durvalumab after four cycles of standard 1st line treatment (Experimental): Study treatment (olaparib and durvalumab) starts with the initiation of maintenance therapy and is administered at a 28-day cycle until progression, unacceptable toxicity, or discontinuation for other reasons.
  Induction therapy (four cycles of carboplatin/cisplatin, etoposide, durvalumab (the administration of one induction cycle without durvalumab is permitted)) is administered as part of standard of care.
  Interventions: Drug: Durvalumab; Drug: Olaparib

INTERVENTIONS:
Drug: Durvalumab — 1500 mg i.v. Q4W
  Other Names: MEDI4736; IMFINZI
Drug: Olaparib — 300 mg BID orally
  Other Names: AZD2281; LYNPARZA

SUMMARY:
Maintenance durvalumab (MEDI4736) and olaparib (AZD2281) after standard 1st line treatment (carboplatin/ cisplatin, etoposide, durvalumab) in HRD positive extensive disease (ED) small-cell lung cancer (SCLC)

ELIGIBILITY:
Inclusion Criteria Pre-Screening:

* Newly diagnosed, histologically documented advanced or metastatic small-cell lung cancer (UICC stage III which is not amenable to curative radiochemotherapy or stage IV). [...]
* Either de novo biopsies collected as part of routine clinical practice or archival tumor samples (taken ≤6 months prior to screening) are acceptable.
* Planned or ongoing treatment with carboplatin/cisplatin, etoposide, durvalumab as 1st-line SoC. Pre-screening must begin no later than the start of the 3rd cycle to allow sufficient time for molecular analyses. [...]
* Available radiographic chest and abdominal CT or MRI scans performed up to 42 days before initial first line treatment with carboplatin/cisplatin, etoposide and durvalumab.
* At least one measurable site of disease as defined by RECIST v1.1 criteria.
* [...]

Inclusion Criteria Screening:

* Completed pre-screening with fulfillment of all inclusion and exclusion criteria of pre-screening. Pre-screening must have tested positive for homologous recombination deficiency as defined in this protocol at central testing. [...]
* Patients must not have radiographic or clinic disease progression while on induction therapy and/or prior to start of study treatment.
* Patients must have received 4 cycles (21-day cycles) of induction with carboplatin or cisplatin, etoposide and durvalumab completed within 1 to 14 days prior to initiation of study treatment on C5D1. Patients must have received durvalumab at minimum three times during the four induction cycles.
* Adequate organ and marrow function

Exclusion Criteria Pre-Screening:

* Induction therapy other than carboplatin/cisplatin, etoposide and durvalumab. (The administration of one induction cycle without durvalumab is permitted.)
* Radiographic or clinical evidence of progressive disease.
* Negative HRD result in a previous pre-screening in this trial.
* [...]

Exclusion Criteria Screening:

* Patients with symptomatic uncontrolled central nervous system (CNS) metastases.
* Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* History of leptomeningeal carcinomatosis.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy. Exceptions are:

  1. Alopecia (any Grade)
  2. Vitiligo (any Grade)
  3. Hypothyroidism stable on hormone replacement (Grade ≤2)
  4. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician
  5. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or olaparib may be included only after consultation with the Sponsor.
  6. ...

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately two years (from First patient in (FSI) to Last patient last visit (LSLV))
  PFS according to investigator-assessed RECIST 1.1 from start of maintenance therapy

SECONDARY OUTCOMES:
Incidence, severity and grading of adverse events (AE) and seriouse adverse events (SAE). | Approximately two years (from FSI to LSLV)
  Grading is based on CTCAE Version 5
ORR of maintenance. | Approximately two years (from FSI to LSLV)
  Grading is based on RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Wolf, MD, Principal Investigator — University Hospital Cologne
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No